CLINICAL TRIAL: NCT02226640
Title: Uncovering the 'ORIGINS' of Diabetes
Acronym: ORIGINS
Status: Completed | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: AdventHealth (Other); Sanford-Burnham Medical Research Institute (Other); UCSF Benioff Children's Hospital Oakland (Other); Duke Univeristy Sarah W. Stedman Nutrition & Metabolism Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: TRIMDFH 238153
Record Dates: First submitted 2014-05-16; First posted 2014-08-27 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Urine Fat tissue Muscle Tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Non-Diabetic Lean Athletes: Athletes with a Body Mass Index (BMI) less than or equal to 25 kg/m2.
- Non-Diabetic Lean No Diabetes History: Adults with a BMI < 25 kg/m2 and no family history of diabetes
- Non-Diabetic Lean Yes Diabetes History: Adults with a BMI < 25 kg/m2 and family history of diabetes
- Non-Diabetic Obese: Adults with BMI greater than or equal to 30 kg/m2.
- Non-Diabetic Obese Female PCOS: Female adults with BMI > 30 kg/m2 and Polycystic Ovarian Syndrome (PCOS).
- Diabetic No Medication: Have diabetes and currently receiving no medication or early treatment with one medication. Some participants receiving insulin may also be included in this study
- Diabetic GAD Ab+: Have diabetes with Latent Autoimmune Diabetes in Adults (LADA).
- Diabetic With NASH: Have diabetes with Nonalcoholic Steatohepatitis (NASH), which is chronic liver disease with fat in the liver, inflammation, and damage not associated with drinking alcohol.

SUMMARY:
This is a study to identify different subtypes of type 2 diabetes. The investigators will look for information at the molecular level, which may lead to personalized diagnosis and therapies.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is approaching epidemic prevalence in the US adult population (over 1 in 10 of all US adults over 20). Diabetes is diagnosed based on fasting hyperglycemia, oral glucose intolerance or markers of hyperglycemia such as HbA1c. However, we now recognize that diabetes is a heterogeneous disorder. With the existing overly simplistic diagnostic criteria, treatment failure rates are high for virtually every agent currently in the drug arsenal - including insulin. In the late 1990's oncologists pioneered the use of high-throughput molecular technologies, such as transcriptome profiling and more recently metabolomics to identify discrete sub-classes of cancers that cannot be distinguished histologically or by a small number of biochemical markers. That effort rapidly accelerated the pace of scientific discovery and quickly led to the development of personalized cancer therapeutics. We believe that those cancer efforts provide a roadmap for biomarker discovery and personalized therapy in diabetes. molecular phenotyping (profiling the metabolome, transcriptome, and epigenome) with advanced bioinformatics analysis will identify discrete subtypes of diabetes - ushering in a new era of personalized diagnosis and therapy in diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* HbA1C < 8.0% *
* You have not gained or lost more than 3 kg or 6.6 pounds in the last 8 weeks
* You have not lost more than 10% of your heaviest body weight in your lifetime
* BMI < 25 kg/m2 or > 30 kg/m2
* Women: more than 1 year post-partum
* Have diabetes and are able to maintain accurate and reliable home glucose monitoring logs

Exclusion Criteria:

* Treatment with more than 2 of the following: metformin (Fortamet, Glucophage, Glumetza, Riomet), sulfonylureas (Glucotrol, Diabeta, Glynase, Micronase), Glucagon-like peptide-1 analogs (Byetta) and/or Dipeptidyl peptidase IV inhibitors (Januvia, Onglyza)
* Treatment with long acting Glucagon-like peptide-1 agonists within the last 3 months (i.e. exenatide once weekly)
* Treatment with thiazolidinediones (TZDs) (i.e. Avandia, Actos, Rezulin) within the last 3 months
* Known, untreated thyroid disease or abnormal thyroid function blood test.*
* Known diagnosis of liver disease (except NASH) or elevated liver function blood test
* Known diagnosis of kidney disease or elevated kidney function blood test
* Uncontrolled high blood pressure (BP > 140 systolic or > 90 diastolic)
* Start of or changes in oral contraceptives or hormone replacement therapy within the last 3 months
* Use of drugs or alcohol (> 3 drinks per day) within the last 5 years.
* Uncontrolled psychiatric disease that would interfere with study participation.
* History of cancer within the last 5 years (skin cancers, with the exception of melanoma, may be acceptable)
* History of organ transplant
* History of heart attack within the last 6 months
* Current treatment with blood thinners or antiplatelet medications that cannot be safely stopped for testing procedures
* Current anemia
* History of HIV, active Hepatitis B or C, or Tuberculosis
* Presence of clinically significant abnormalities on electrocardiogram.
* Current smokers (smoking any nicotine or non-nicotine product within the past 3 months)
* Use of any medications known to influence glucose, fat and/or energy metabolism within the last 3 months (e.g., growth hormone therapy, glucocorticoids [steroids], etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Perform 'deep' clinical and molecular phenotyping of 360 adults- Diabetic and Non-Diabetic | up to Day 9
  Phenotyping will include whole body composition (DEXA), substrate metabolism, classic diabetes phenotypes, and detailed molecular phenotyping of circulating mononuclear cells/ plasma, muscle and adipose tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, MD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

REFERENCES:
- [Background] Shoelson SE, Lee J, Yuan M. Inflammation and the IKK beta/I kappa B/NF-kappa B axis in obesity- and diet-induced insulin resistance. Int J Obes Relat Metab Disord. 2003 Dec;27 Suppl 3:S49-52. doi: 10.1038/sj.ijo.0802501. PMID 14704745
- [Background] Reitman ML, Arioglu E, Gavrilova O, Taylor SI. Lipoatrophy revisited. Trends Endocrinol Metab. 2000 Dec;11(10):410-6. doi: 10.1016/s1043-2760(00)00309-x. PMID 11091118
- [Background] Itani SI, Ruderman NB, Schmieder F, Boden G. Lipid-induced insulin resistance in human muscle is associated with changes in diacylglycerol, protein kinase C, and IkappaB-alpha. Diabetes. 2002 Jul;51(7):2005-11. doi: 10.2337/diabetes.51.7.2005. PMID 12086926
- [Background] Moro C, Bajpeyi S, Smith SR. Determinants of intramyocellular triglyceride turnover: implications for insulin sensitivity. Am J Physiol Endocrinol Metab. 2008 Feb;294(2):E203-13. doi: 10.1152/ajpendo.00624.2007. Epub 2007 Nov 14. PMID 18003718
- [Background] Kelley DE, He J, Menshikova EV, Ritov VB. Dysfunction of mitochondria in human skeletal muscle in type 2 diabetes. Diabetes. 2002 Oct;51(10):2944-50. doi: 10.2337/diabetes.51.10.2944. PMID 12351431
- [Background] Ritov VB, Menshikova EV, Azuma K, Wood R, Toledo FG, Goodpaster BH, Ruderman NB, Kelley DE. Deficiency of electron transport chain in human skeletal muscle mitochondria in type 2 diabetes mellitus and obesity. Am J Physiol Endocrinol Metab. 2010 Jan;298(1):E49-58. doi: 10.1152/ajpendo.00317.2009. Epub 2009 Nov 3. PMID 19887598
- [Background] Alizadeh AA, Eisen MB, Davis RE, Ma C, Lossos IS, Rosenwald A, Boldrick JC, Sabet H, Tran T, Yu X, Powell JI, Yang L, Marti GE, Moore T, Hudson J Jr, Lu L, Lewis DB, Tibshirani R, Sherlock G, Chan WC, Greiner TC, Weisenburger DD, Armitage JO, Warnke R, Levy R, Wilson W, Grever MR, Byrd JC, Botstein D, Brown PO, Staudt LM. Distinct types of diffuse large B-cell lymphoma identified by gene expression profiling. Nature. 2000 Feb 3;403(6769):503-11. doi: 10.1038/35000501. PMID 10676951
- [Background] Sreekumar A, Poisson LM, Rajendiran TM, Khan AP, Cao Q, Yu J, Laxman B, Mehra R, Lonigro RJ, Li Y, Nyati MK, Ahsan A, Kalyana-Sundaram S, Han B, Cao X, Byun J, Omenn GS, Ghosh D, Pennathur S, Alexander DC, Berger A, Shuster JR, Wei JT, Varambally S, Beecher C, Chinnaiyan AM. Metabolomic profiles delineate potential role for sarcosine in prostate cancer progression. Nature. 2009 Feb 12;457(7231):910-4. doi: 10.1038/nature07762. PMID 19212411
- [Background] van't Veer LJ, Bernards R. Enabling personalized cancer medicine through analysis of gene-expression patterns. Nature. 2008 Apr 3;452(7187):564-70. doi: 10.1038/nature06915. PMID 18385730
- [Background] Wang S, Sparks LM, Xie H, Greenway FL, de Jonge L, Smith SR. Subtyping obesity with microarrays: implications for the diagnosis and treatment of obesity. Int J Obes (Lond). 2009 Apr;33(4):481-9. doi: 10.1038/ijo.2008.277. Epub 2009 Feb 3. PMID 19188926
- [Background] Ptitsyn A, Hulver M, Cefalu W, York D, Smith SR. Unsupervised clustering of gene expression data points at hypoxia as possible trigger for metabolic syndrome. BMC Genomics. 2006 Dec 19;7:318. doi: 10.1186/1471-2164-7-318. PMID 17178004
- [Background] Naik RG, Brooks-Worrell BM, Palmer JP. Latent autoimmune diabetes in adults. J Clin Endocrinol Metab. 2009 Dec;94(12):4635-44. doi: 10.1210/jc.2009-1120. Epub 2009 Oct 16. PMID 19837918
- [Background] West M, Blanchette C, Dressman H, Huang E, Ishida S, Spang R, Zuzan H, Olson JA Jr, Marks JR, Nevins JR. Predicting the clinical status of human breast cancer by using gene expression profiles. Proc Natl Acad Sci U S A. 2001 Sep 25;98(20):11462-7. doi: 10.1073/pnas.201162998. Epub 2001 Sep 18. PMID 11562467
- [Background] Sorlie T. Molecular portraits of breast cancer: tumour subtypes as distinct disease entities. Eur J Cancer. 2004 Dec;40(18):2667-75. doi: 10.1016/j.ejca.2004.08.021. PMID 15571950
- [Background] Sorlie T. Introducing molecular subtyping of breast cancer into the clinic? J Clin Oncol. 2009 Mar 10;27(8):1153-4. doi: 10.1200/JCO.2008.20.6276. Epub 2009 Feb 9. No abstract available. PMID 19204193
- [Background] Perou CM, Sorlie T, Eisen MB, van de Rijn M, Jeffrey SS, Rees CA, Pollack JR, Ross DT, Johnsen H, Akslen LA, Fluge O, Pergamenschikov A, Williams C, Zhu SX, Lonning PE, Borresen-Dale AL, Brown PO, Botstein D. Molecular portraits of human breast tumours. Nature. 2000 Aug 17;406(6797):747-52. doi: 10.1038/35021093. PMID 10963602
- [Background] Mutch DM, Temanni MR, Henegar C, Combes F, Pelloux V, Holst C, Sorensen TI, Astrup A, Martinez JA, Saris WH, Viguerie N, Langin D, Zucker JD, Clement K. Adipose gene expression prior to weight loss can differentiate and weakly predict dietary responders. PLoS One. 2007 Dec 19;2(12):e1344. doi: 10.1371/journal.pone.0001344. PMID 18094752
- [Background] Henry RR, Abrams L, Nikoulina S, Ciaraldi TP. Insulin action and glucose metabolism in nondiabetic control and NIDDM subjects. Comparison using human skeletal muscle cell cultures. Diabetes. 1995 Aug;44(8):936-46. doi: 10.2337/diab.44.8.936. PMID 7622000
- [Background] Ukropcova B, McNeil M, Sereda O, de Jonge L, Xie H, Bray GA, Smith SR. Dynamic changes in fat oxidation in human primary myocytes mirror metabolic characteristics of the donor. J Clin Invest. 2005 Jul;115(7):1934-41. doi: 10.1172/JCI24332. PMID 16007256
- [Background] Aagaard-Tillery KM, Grove K, Bishop J, Ke X, Fu Q, McKnight R, Lane RH. Developmental origins of disease and determinants of chromatin structure: maternal diet modifies the primate fetal epigenome. J Mol Endocrinol. 2008 Aug;41(2):91-102. doi: 10.1677/JME-08-0025. Epub 2008 May 30. PMID 18515302
- [Background] Cox J, Williams S, Grove K, Lane RH, Aagaard-Tillery KM. A maternal high-fat diet is accompanied by alterations in the fetal primate metabolome. Am J Obstet Gynecol. 2009 Sep;201(3):281.e1-9. doi: 10.1016/j.ajog.2009.06.041. PMID 19733280
- [Background] Barker DJ, Gluckman PD, Godfrey KM, Harding JE, Owens JA, Robinson JS. Fetal nutrition and cardiovascular disease in adult life. Lancet. 1993 Apr 10;341(8850):938-41. doi: 10.1016/0140-6736(93)91224-a. PMID 8096277
- [Background] Barker DJ, Hales CN, Fall CH, Osmond C, Phipps K, Clark PM. Type 2 (non-insulin-dependent) diabetes mellitus, hypertension and hyperlipidaemia (syndrome X): relation to reduced fetal growth. Diabetologia. 1993 Jan;36(1):62-7. doi: 10.1007/BF00399095. PMID 8436255
- [Background] Barres R, Osler ME, Yan J, Rune A, Fritz T, Caidahl K, Krook A, Zierath JR. Non-CpG methylation of the PGC-1alpha promoter through DNMT3B controls mitochondrial density. Cell Metab. 2009 Sep;10(3):189-98. doi: 10.1016/j.cmet.2009.07.011. PMID 19723495
- [Background] Freda PU, Shen W, Reyes-Vidal CM, Geer EB, Arias-Mendoza F, Gallagher D, Heymsfield SB. Skeletal muscle mass in acromegaly assessed by magnetic resonance imaging and dual-photon x-ray absorptiometry. J Clin Endocrinol Metab. 2009 Aug;94(8):2880-6. doi: 10.1210/jc.2009-0026. Epub 2009 Jun 2. PMID 19491226
- [Background] Welch S, Gebhart SS, Bergman RN, Phillips LS. Minimal model analysis of intravenous glucose tolerance test-derived insulin sensitivity in diabetic subjects. J Clin Endocrinol Metab. 1990 Dec;71(6):1508-18. doi: 10.1210/jcem-71-6-1508. PMID 2229309
- [Background] Bergman RN, Ider YZ, Bowden CR, Cobelli C. Quantitative estimation of insulin sensitivity. Am J Physiol. 1979 Jun;236(6):E667-77. doi: 10.1152/ajpendo.1979.236.6.E667. PMID 443421
- [Background] Elia M, Livesey G. Energy expenditure and fuel selection in biological systems: the theory and practice of calculations based on indirect calorimetry and tracer methods. World Rev Nutr Diet. 1992;70:68-131. doi: 10.1159/000421672. No abstract available. PMID 1292242
- [Background] Brody DL, Magnoni S, Schwetye KE, Spinner ML, Esparza TJ, Stocchetti N, Zipfel GJ, Holtzman DM. Amyloid-beta dynamics correlate with neurological status in the injured human brain. Science. 2008 Aug 29;321(5893):1221-4. doi: 10.1126/science.1161591. PMID 18755980
- [Background] Smith, S.R., Martin, C., Katzmarzyk, P. & Church, T. Obesity and Diabetes: Implications for Management. in 2009 Educational Review Manual in Endocrinology FOCUS: Diabetes (ed. Kendall, D.M.) (Castle Connolly Graduate Medical Publishing, New York, NY 2009).
- [Derived] Divoux A, Eroshkin A, Erdos E, Sandor K, Osborne TF, Smith SR. DNA Methylation as a Marker of Body Shape in Premenopausal Women. Front Genet. 2021 Jul 29;12:709342. doi: 10.3389/fgene.2021.709342. eCollection 2021. PMID 34394195
- [Derived] Pachori AS, Madan M, Nunez Lopez YO, Yi F, Meyer C, Seyhan AA. Reduced skeletal muscle secreted frizzled-related protein 3 is associated with inflammation and insulin resistance. Obesity (Silver Spring). 2017 Apr;25(4):697-703. doi: 10.1002/oby.21787. Epub 2017 Feb 27. PMID 28240822
- See also: Florida Hospital Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org